CLINICAL TRIAL: NCT05763771
Title: Smartphone-delivered Scheduled Smoking With Compliance Facilitation as an Adjunct Cessation Therapy: a Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-0772; NCI-2023-01983 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-23; First posted 2023-03-10 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): Participants will use the app for 4 weeks, during which participants will follow a smoking schedule on the app to help you reduce your cigarette consumption
  Interventions: Behavioral: Smart Phone App; Other: NIcotine Patches
- Part 2 (Experimental): Participants will also use the app for the duration of the study (about 3 months).
  Participants will be asked to record your smoking using the app and complete online surveys
  Interventions: Behavioral: Smart Phone App; Other: NIcotine Patches

INTERVENTIONS:
Behavioral: Smart Phone App — Collection of data
Other: NIcotine Patches — Place on the skin

SUMMARY:
To collect user experience data for a smartphone app that is designed to help people reduce or quit smoking and to learn if the app, combined with nicotine patches, can help people quit smoking.

DETAILED DESCRIPTION:
Objectives:

We propose to develop a mobile smoking intervention termed COmpliance-facilitated Scheduled Smoking Reduction (COSSR) delivered as a smartphone app. Through the proposed research as a pilot study, we want to identify the effect size of the proposed COSSR

intervention. We will pursue the following aims:

Aim 1:

Develop the COSSR app and evaluate the app's usability. In this aim, our first objective is to develop the COSSR app, and our second objective is to evaluate the app's usability, making sure that our app's core features are working, such as generating personalized smoking schedules, recording smoking, and taking carbon monoxide (CO) measures using the portable CO devices. We will recruit 15 participants from across the state of Texas to test our app for 4 weeks.

Aim 2:

Evaluate COSSR's preliminary effects on smoking cessation. In this aim, we will recruit participants (n=60) remotely from across the entire state of Texas to evaluate COSSR's effects on smoking cessation. Participants will be randomly assigned to either the control or the COSSR group. Both groups include the usual care treatment (self-help material and nicotine patches). In the COSSR group, they will use the app to reduce their smoking before quitting, and use 3-week pre-cessation nicotine patches.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 years old or older

* Smoking: an average of 10 or more cigarettes, little cigars, or cigarillos combined per day within the past 30 days preceding the phone screen
* Expired carbon monoxide (CO): > 6 ppm
* Can install and run the study app on their Android smartphone, or agree to use the study smartphone loaned from the research team
* Agree to return the study smartphone if the participant loans one from the research team
* Willing to reduce smoking (Aim 1)
* Seeking smoking cessation treatment (Aim 2)
* Fluency in spoken and written English
* Agree to be treated via telehealth (live audio-video conference and phone) and to be contacted via text and/or email
* Provide informed consent and agree to all assessments and study procedures
* Willing to refrain from the use of other nicotine/tobacco products for the duration of the study
* Willing to refrain from the use of marijuana, prescription medications not prescribed to the participant, and illegal drugs

Exclusion Criteria:

* Taking psychotropic, anticonvulsive, or narcotic medication
* Meet criteria for a current major depressive episode or suicidality according to the PHQ (indicated by a score of 10 or higher).
* Involved in current and imminent (within the next 45 days) smoking cessation activity
* Women who are pregnant or breastfeeding
* Shares the same address as a currently enrolled participant
* Unwilling to use or allergic to nicotine patches (Aim 2)
* Considered by the investigator to be an unsuitable or unstable candidate, such as those who appear to have cognitive impairment, and those who reside in a shelter, group/recovery facility, or treatment facility
* Any plans to move out of the state in the next 6 months
* Using marijuana, prescription medications not prescribed to the participant, and illegal drugs on a daily basis
* Have experienced abnormal heart rhythms or cardiovascular disease, such as stroke, chest pain, and heart attack, in the last month (Aim 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Application (App) Usability Questionnaire | through completion of study; an average of 1 year.
  Scale Scores (1-5) 1-strongly disagree, 2-disagree, 3-neither disagree nor agree, 4-agree and 5-strongly agree

CONTACTS AND LOCATIONS:
Overall Officials: Yong Cui, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2024-09-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT05763771/ICF_001.pdf